CLINICAL TRIAL: NCT06506760
Title: The Impact of Immersive Virtual Reality Therapy on Psychological and Functional Status in Female Patients Undergoing Inpatient Rehabilitation Following Hip Arthroplasty: A Randomized Controlled Pilot Study
Brief Title: Immersive VR for Female Orthopaedic Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Wroclaw Medical University (Other); Jan Dlugosz University in Czestochowa (Other)
Responsible Party: Principal Investigator, Joanna Szczepańska-Gieracha, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRortov2
Record Dates: First submitted 2024-07-09; First posted 2024-07-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthropathy
Keywords: virtual reality; arthroplasty; women; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality Therapy (Experimental): Conventional orthopedic rehabilitation supplemented by VR therapy
  Interventions: Behavioral: Immersive Virtual Reality Therapy
- Conventional rehabilitation (Active Comparator): Conventional orthopedic rehabilitation
  Interventions: Behavioral: Immersive Virtual Reality Therapy; Behavioral: Conventional rehabilitation

INTERVENTIONS:
Behavioral: Immersive Virtual Reality Therapy — 8 sessions of VR therapy over 4 weeks (each of them 20 minutes long).
  As a virtual reality source, VRTierOne device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion VR therapy provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach. The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the therapist tells the patient a symbolic story about his/her situation.
Behavioral: Conventional rehabilitation — Four weeks of conventional rehabilitation including:
  Two hours of kinesiotherapy (120 minutes, including gait training). Thirty minutes of ergotherapy. Three physical therapy procedures (i.e. laser therapy, magnetic therapy, electrotherapy) tailored to individual ailments and needs.
  Arms: Conventional rehabilitation

SUMMARY:
This study compares the effects of cardiological rehabilitation enhanced with virtual reality (VR) versus conventional rehabilitation methods. It assesses the impact on both psychological parameters (including depression, stress, anxiety, and kinesiophobia) and physiological and functional parameters of cardiology patients. The aim is to analyze the efficacy and benefits of VR-supported rehabilitation in improving patients' mental and physical health compared to traditional methods.

DETAILED DESCRIPTION:
The study will involve elderly female patients aged 60 and above who present sequentially at the Rehabilitation Department of St. Hedwig of Silesia Hospital in Trzebnica (Poland) within three months following hip joint arthroplasty surgery. Participants will be randomly assigned to one of two groups: Group A, the Virtual Reality Group, will receive 8 therapy sessions, with two sessions per week; Group B, the Control Group, will undergo conventional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals who have recently undergone hip joint arthroplasty surgeries aged 60 years and above.

Exclusion Criteria:

* cognitive impairments that prevent independent completion of research questionnaires
* reported consciousness disorders
* bipolar affective disorder and other serious mental disorders in the patient's medical history
* use of psychoactive drugs
* ongoing psychiatric treatment or individual psychological therapy
* contraindications to Virtual Reality such as epilepsy, vertigo, serious vision disorders
* functional status preventing independent movement (orthopedic aids are allowed, e.g., crutches, walker)
* refusal to participate in the study at any stage

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline and 4 weeks
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms.

SECONDARY OUTCOMES:
Perceived Stress Scale | Baseline and 4 weeks
  The Perceived Stress Scale (PSS-10) is a ten-item scale that assesses the level of stress perceived by an individual in the last month. The questions are general in nature and fairly free of content specific to any subpopulation group. The items are designed to tap into how unpredictable, uncontrollable, and overloaded respondents find their lives to be. The scores range from 0 to 40, with higher scores indicating higher perceived stress. The Perceived Stress Scale will be administered at the beginning and after four weeks of treatment.
Generalized Self-Efficacy Scale | Baseline and 4 weeks
  The Generalized Self-Efficacy Scale (GSES) is a ten-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. The scale measures the belief in one's competence to cope with a broad range of stressful or challenging demands. The score ranges from 10 to 40, with a higher score indicating a greater sense of self-efficacy. The Generalized Self-Efficacy Scale will be applied at the beginning and after four weeks of treatment.
Barthel Index | Baseline and 4 weeks
  The Barthel Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing activities of daily living and mobility. Scores range from 0 to 100, with higher scores associated with a greater likelihood of being able to live at home with a degree of independence following discharge from the hospital. The Barthel Index will be administered at the beginning and after four weeks of treatment.
Rivermead Mobility Index | Baseline and 4 weeks
  The Rivermead Mobility Index (RMI) was developed from the Rivermead Motor Assessment Gross Function subscale as a means to quantify mobility disability. It is composed of 14 items representing different mobility tasks, ranging from turning over in bed to running. Each item is scored as 'unable' (0) or 'able' (1), leading to a maximum score of 14, which indicates full mobility. The Rivermead Mobility Index will be administered at the beginning and after four weeks of treatment.
Tinetti's Short Scale | Baseline and 4 weeks
  Tinetti's Short Scale for fall risk assessment is a shortened version of Performance-Oriented Mobility Assessment (POMA). It is easily administered test that measures a patient's gait and balance. The test is scored on the patient's ability to perform following tasks: Change from sitting to standing, Immobilization in standing position for 5 seconds, Passing 3 meters, Turn of 180 degrees, Keeping a sitting position. Each task is rated in 3-point Likert scale. The scales rage from 0-15, with the higher scores indicate better functional mobility.
Short Physical Performance Battery | Baseline and 4 weeks
  The Short Physical Performance Battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It provides a composite score ranging from 0 (worst performance) to 12 (best performance), offering a global assessment of physical functioning in older individuals. The SPPB will be administered at the beginning and after four weeks of treatment.
Perception of Stress Questionnaire | Baseline and 4 weeks
  The Perception of Stress Questionnaire (PSQ) was created by Plopa and Makarowski. It is a 27-item scale scoring from 1 to 5 points for each item, where 21 items examine the level of stress in the areas of emotional tension, external stress and intrapsychic stress, and six items refer to the lie scale. The global scoring for the perception of stress ranges from 21 to 105, with a cut-off point of 60 for an elevated level of perceived stress. Higher scores indicate higher stress perception.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Mazurek, PhD, Principal Investigator — Wroclaw Medical University; Joanna Szczepańska-Gieracha, Professor, Study Chair — Wrocław University of Health and Sport Sciences; Robert Gajda, PhD, Study Chair — Gajda-Med District Hospital in Pułtusk
Locations (1):
- St. Hedwig of Silesia Hospital, Trzebnica, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cieslik B, Mazurek J, Rutkowski S, Kiper P, Turolla A, Szczepanska-Gieracha J. Virtual reality in psychiatric disorders: A systematic review of reviews. Complement Ther Med. 2020 Aug;52:102480. doi: 10.1016/j.ctim.2020.102480. Epub 2020 Jun 9. PMID 32951730
- [Background] Szczepanska-Gieracha J, Cieslik B, Rutkowski S, Kiper P, Turolla A. What can virtual reality offer to stroke patients? A narrative review of the literature. NeuroRehabilitation. 2020;47(2):109-120. doi: 10.3233/NRE-203209. PMID 32741792
- [Background] Szczepanska-Gieracha J, Jozwik S, Cieslik B, Mazurek J, Gajda R. Immersive Virtual Reality Therapy as a Support for Cardiac Rehabilitation: A Pilot Randomized-Controlled Trial. Cyberpsychol Behav Soc Netw. 2021 Aug;24(8):543-549. doi: 10.1089/cyber.2020.0297. Epub 2021 Feb 11. PMID 33577375
- [Background] Wrzeciono A, Cieslik B, Kiper P, Szczepanska-Gieracha J, Gajda R. Exploratory analysis of the effectiveness of virtual reality in cardiovascular rehabilitation. Sci Rep. 2024 Jan 2;14(1):281. doi: 10.1038/s41598-023-50788-9. PMID 38168468
- [Background] Mazurek J, Cieslik B, Wrzeciono A, Gajda R, Szczepanska-Gieracha J. Immersive Virtual Reality Therapy Is Supportive for Orthopedic Rehabilitation among the Elderly: A Randomized Controlled Trial. J Clin Med. 2023 Dec 14;12(24):7681. doi: 10.3390/jcm12247681. PMID 38137750